CLINICAL TRIAL: NCT04814251
Title: A Prospective and Multicentric Cohort Study Evaluating the Complications of Portal Vein Thrombosis in Patients With Locally Advanced Pancreatic Cancer : THROMPAN
Brief Title: Portal Vein Thrombosis Associated With Unresectable Pancreatic Cancers : a Prospective Multicentric Cohort Study
Acronym: THROMPAN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: THROMPAN
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observationnal cohort — data collection

SUMMARY:
Little is known concerning the management of portal vein thrombosis (PVT) in digestive cancers other than hepato-cellular carcinoma (HCC). The use of anticoagulant treatment (ACT), screening of oesophageal varices (OV) and oesogatric varices (OGV), and primary prophylaxis of OV (treatment with beta-blocker (BB) and / or OV ligation) if necessary are not clearly defined. The autopsy series by Ogren et al. (World J Gastroenterol. 2006) found an incidence of PVT in cancer patients of 1%, with 44% of digestive cancers other than HCC as a common etiology, mostly pancreatic adenocarcinoma (42%).

We reported a retrospective French study that included 118 patients with digestive cancers other than HCC, including 50% locally advanced or metastatic pancreatic adenocarcinoma, with PVT complications. A total of 38% of patients had radiological signs of portal hypertension (PHT) and 51% had ACT. Only 1% of patients were screened for VO (n = 7). In addition, 19% (n = 22) presented gastrointestinal bleeding. Among the causes of death, 17% (n = 12) were due to gastrointestinal bleeding. Overall survival (OS) was statistically associated with a metastatic disease (HR = 2.83 [95% CI 1.47-5.43], p <0.01) and gastrointestinal bleeding (HR = 1.68 [95% CI 1.01-2.78], p = 0.04).

Bleeding complications from PHT are not uncommon in patients with digestive cancer, especially in patients with pancreatic cancer with PVT; but above all they can be responsible for death. No data existed before our first study (Regnault et al. Dig Liv Dis 2018). However, these data must be validated in a prospective multicentric study with standardized follow-up. In order to obtain precise and homogeneous data, we have chosen to target pancreatic cancers as these tumors are the most common causes of PVT.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic adenocarcinoma proven histologically or cytologically in favor of pancreatic adenocarcinoma
* Mesurable disease according to RECIST 1.1 criteria or non measurable disease
* Metastatic disease (synchronous or metachronous) or locally advanced / borderline deemed unresectable and / or patient inoperable due to his co-morbidities and / or local recurrence after surgery
* Thrombosis of the main portal vein and/or of one of its branches (endo-luminal defect on the injected CTscan) of cruoric or tumoral origin or circumferential stenosis of the portal vein trunk, the spleno-mesaraic confluence or one of its venous branches with or without signs of portal hypertension on CTscan and / or upper GIendoscopy

Exclusion Criteria:

* - Post-surgical portal vein thrombosis and / or in patients considered in remission
* Non-adenocarcinomatous pancreatic tumor (endocrine, etc.)

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients followed for unresectable pancreatic adenocarcinoma with portal vein thrombosis or portal hypertension with scan evidence (splenomegaly and/or portosystemic shunts).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of digestive and non-digestive bleeding | 18 months
  Hematemesis, melena and / or rectal bleeding Hematuria, intra-abdominal, intracranial bleeding and / or other bleeding considered clinically relevant by the investigators

SECONDARY OUTCOMES:
Screening rate of oesophageal varices by upper gastriintestinal endoscopy, | 18 months
Detection rate of oesophageal varices | 18 months
Rate of primary prophylaxis of oesophageal varices | 18 months
Rate of secondary prophylaxis of oesophageal varices | 18 months
Rate of anticoagulant treatment use | 18 months
Portal hypertension related death, predictive factors of gastrointestinal bleeding and overall survival. | 18 months

IPD SHARING:
Plan to Share IPD: No